CLINICAL TRIAL: NCT06009575
Title: Local Culture-Based Nutrition Education Intervention on Iron Supplement Tablets (IST) Consumption Compliance in Female Adolescents at Ogan Komering Ilir Regency: A Quasi-Experimental Protocol Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Anita Rahmiwati, Dr, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: US
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Anemia; Iron Deficiency Anemia
Keywords: anemia; Iron Supplement Tablets
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Dietary Supplement: Iron Supplement Tablets
- control group (Active Comparator)
  Interventions: Dietary Supplement: Iron Supplement Tablets

INTERVENTIONS:
Dietary Supplement: Iron Supplement Tablets — The intervention group received IST and local culture-based nutrition education

SUMMARY:
The goal of this clinical trial is to test the impact of a local culture-based nutritional education intervention on IST consumption compliance among female adolescents in the Ogan Komering Ilir Regency. The main questions it aims to answer are:

a To identify information for the development of a local culture-based nutrition education model and to build a ready-to-implement local culture-based nutrition education model.

b. To evaluate the implementation of the Anemia Prevention and Control Program among female adolescents in Ogan Komering Ilir Regency.

c. To test the impact of the local culture-based nutrition education model on the improvement of knowledge, attitude, and IST consumption compliance among female adolescents.

Participants will received IST and local culture-based nutrition education. Researchers will compare control group received IST as the Ministry of Health's program for the prevention of anemia with a subsidy for providing IST

ELIGIBILITY:
Inclusion Criteria:

* public schools have received the IST program from the government, and the distance between schools is at least 10 kilometers
* students enrolled in grade 11, age range 15-17 years, menstruating, owning a smartphone, having an Instagram account, and obtaining parental approval to participate in this study

Exclusion Criteria:

* schools that are currently the object of another study and are difficult to reach (remote areas)
* students who have a BMI value≤ -3 SD and do not watch complete educational videos for the sample in the intervention group

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Educational Intervention | 12 Weeks
  The local culture to be used was based on the results of a qualitative study conducted prior to the intervention, where Kelakar Betok is the local culture preferred by female adolescents, used as a means of nutrition education. Subsequently, the social media used in nutrition education publicity is Instagram. Nutrition education is provided in the form of educational videos based on local culture broadcasted through the Instagram account @remaja.bebasanemia.
Iron Supplement Tablet (IST) Administration | 16 Weeks
  The IST used as an intervention consists of IST containing 60 mg FeSO4 and 400 mcg of folic acid, which is a government program. The program policy for administering IST to female adolescents is carried out once a week in the year, which was given in a blanket approach. This supplementation was carried out at educational institutions. The schools that receive iron tablets are Junior High Schools and Senior High Schools

CONTACTS AND LOCATIONS:
Locations (1):
- Anita Rahmiwati, Palembang, South Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan (SAP)